CLINICAL TRIAL: NCT04233697
Title: Phase 1B Study of the PI3K Inhibitor Copanlisib in Combination With Romidepsin in the Treatment of Patients With Relapsed or Refractory Mature T-cell Lymphoma
Brief Title: Copanlisib in Combination With Romidepsin in Patients With Relapsed or Refractory Mature T-cell Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: Columbia University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAR5207
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Lymphoma, T-Cell
Keywords: Hodgkin lymphoma (HL); non-Hodgkin lymphoma (NHL); Copanlisib; Romidepsin
MeSH Terms: conditions — Lymphoma, T-Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — copanlisib; romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Copanlisib and Romidepsin (Experimental): Copanlisib and romidepsin will be both administered via IV (through a vein in arm) on days 1, 8, and 15 every 28 days, also called a "cycle".
  Interventions: Drug: Copanlisib; Drug: Romidepsin

INTERVENTIONS:
Drug: Copanlisib — Novel, pan-class phosphatidylinositol 3-kinase (PI3K) inhibitor with potent activity against both the δ and α isoforms9. Copanlisib has been evaluated for the treatment of a wide variety of malignancies, including lymphoma, either as a single agent or in combination with other investigational agents.
  Other Names: Aliqopa; 80-6946
Drug: Romidepsin — Indicated for treatment of cutaneous T-cell lymphoma (CTCL) in patients who have received at least one prior systemic therapy.
  Other Names: Istodax

SUMMARY:
This is an open label, Phase IB dose-escalation study of the PI3K inhibitor copanlisib in combination with romidepsin in patients with relapsed or refractory (R/R) non-Hodgkin lymphoma (NHL) or Hodgkin lymphoma (HL).

The primary objective of the phase I study is to determine the maximum tolerated dose (MTD), recommended phase 2 dose (RP2D), and dose limiting toxicities (DLTs) of the combination of copanlisib and romidepsin in patients with R/R, NHL or HL.

DETAILED DESCRIPTION:
The non-Hodgkin lymphomas (NHL) represent 4-5% of all new cancer cases, and is the seventh leading cause of cancer death. In 2015, there were an estimated 71,850 cases in the United States, and approximately 19,790 deaths. An evaluation of the distribution of NHL sub-types was performed on 114,548 cases of lymphoid neoplasms diagnosed between 1992-2001 and reported to the Surveillance Epidemiology and End Results (SEER) registry. Of all NHL, 87,666 were B-cell lymphoid neoplasms, and 6,228 were considered T/Natural Killer (NK) cell neoplasms.

The peripheral T-cell lymphomas (PTCL) are a heterogeneous group of aggressive lymphoid neoplasms and account for 10-15% of all newly diagnosed cases of NHL. The current prevalence of PTCL in the United States is estimated to be approximately 9,500 patients. PTCL-Not Otherwise Specified (NOS), a nodal subtype, is the most common T-cell lymphoma in the United States and Europe. PTCL is associated with a significantly worse prognosis compared to its B-cell counterparts. Treatment options for patients with relapsed/refractory (R/R) PTCL have been limited. The addition of novel drugs to conventional chemotherapy has largely proven unsuccessful. Since 2009, new drugs have entered the therapeutic field for patients with R/R PTCL.

Pralatrexate was the first drug approved for patients with R/R PTCL. Other drugs approved for patients with R/R PTCL include romidepsin and belinostat. These agents appear to exhibit lineage-specific activity in PTCL. Over the past few years, the investigators have focused on exploring rational combinations of these T-cell active agents in an effort to develop novel treatment platforms. Early clinical studies of these combinations have shown very promising activity.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Be ≥18 years of age on day of signing informed consent.
* Have measurable disease based on the Lugano Criteria.
* Phase I: patient must have histologically confirmed R/R NHL or HL (defined by World Health Organization (WHO) criteria).
* Expansion phase: patients must have histologically confirmed R/R mature T-cell lymphoma (defined by WHO criteria).
* Patient must have received at least two prior lines of therapy prior to enrollment in this study.
* Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Left Ventricular Ejection Fraction (LVEF) > 50%.
* Demonstrate adequate organ function. All screening labs should be performed within 10 days of treatment initiation. The following treatments are prohibited: (a) Chemotherapy, monoclonal antibody within 4 weeks; (b) radiotherapy within 2 weeks prior to entering the study; (c) systemic steroids that have not been stabilized (≥ 5 days) to the equivalent of ≤10 mg/day prednisone prior to the start of the study drugs; (d) other concurrent investigational agents within 4 weeks prior to entering the study; (e) use of copanlisib or romidepsin within the past 3 months.
* Patients that have not recovered from adverse events due to chemotherapy agents administered more than 4 weeks earlier.
* Hypersensitivity to copanlisib or romidepsin or any of its excipients.
* Patients that received major surgery and have not recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Patients with active, clinically serious infections > CTCAE Grade 2.
* Patients with Cytomegalovirus (CMV) PCR positive at baseline.
* Patients with active infections including: active tuberculosis (TB), Hepatitis B (e.g., HBsAg reactive), Hepatitis C, Hepatitis A.
* Patients with uncontrolled inter-current illness (e.g. pneumonia).
* Patients with known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies
* Adequate Contraception.

Exclusion Criteria:

* The following treatments are prohibited: (a) Chemotherapy, monoclonal antibody within 4 weeks; (b) radiotherapy within 2 weeks prior to entering the study; (c) systemic steroids that have not been stabilized (≥ 5 days) to the equivalent of ≤10 mg/day prednisone prior to the start of the study drugs; (d) other concurrent investigational agents within 4 weeks prior to entering the study; (e) use of copanlisib or romidepsin within the past 3 months.
* Patients that have not recovered from adverse events due to chemotherapy agents administered more than 4 weeks earlier.
* Hypersensitivity to copanlisib or romidepsin or any of its excipients.
* Patients that received major surgery and have not recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Patients with active, clinically serious infections > CTCAE Grade 2.
* Patients with CMV PCR positive at baseline.
* Patients with active infections including: active TB (Mycobacterium Tuberculosis), Hepatitis B (e.g., HBsAg reactive), Hepatitis C (e.g., HCV RNA [qualitative] is detected), Hepatitis A.
* Patients with uncontrolled inter-current illness (e.g. pneumonia).
* Patients with known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies The following treatments are prohibited: (a) Chemotherapy, monoclonal antibody within 4 weeks; (b) radiotherapy within 2 weeks prior to entering the study; (c) systemic steroids that have not been stabilized (≥ 5 days) to the equivalent of ≤10 mg/day prednisone prior to the start of the study drugs; (d) other concurrent investigational agents within 4 weeks prior to entering the study; (e) use of copanlisib or romidepsin within the past 3 months.
* Patients that have not recovered from adverse events due to chemotherapy agents administered more than 4 weeks earlier.
* Hypersensitivity to copanlisib or romidepsin or any of its excipients.
* Patients that received major surgery and have not recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Patients with active, clinically serious infections > CTCAE Grade 2.
* Patients with CMV PCR positive at baseline.
* Patients with active infections including: active TB (Mycobacterium Tuberculosis), Hepatitis B (e.g., HBsAg reactive), Hepatitis C (e.g., HCV RNA [qualitative] is detected), Hepatitis A.
* Patients with uncontrolled inter-current illness (e.g. pneumonia).
* Patients with known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies
* Patients with known active concurrent malignancy (except non-melanoma skin cancer, prostatic intraepithelial neoplasia, or carcinoma in situ of the cervix). If there is a history of prior malignancy, the patient must be disease-free for ≥ 3 years.
* Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis and/or known lymphomatous involvement of the central nervous system.
* Evidence of active non-infectious pneumonitis (NIP).
* History of concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator).
* Patients with an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Of note, replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed for patient on study.
* Uncontrolled Type I or II diabetes mellitus as deemed appropriate by the investigator (suggested guidelines for uncontrolled diabetes: HbA1c> 8.5%).
* Uncontrolled hypertension, i.e., blood pressure (BP) of ≥ 150/90; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria.
* Concomitant use of CYP3A4 inhibitors.
* Congenital long QT syndrome and/or QTc interval ≥ 500 milliseconds.
* Patients taking drugs leading to significant QT prolongation.
* Any cardiac arrhythmia requiring an anti-arrhythmic medication, with the exception of stable doses of beta-blockers.
* Myocardial infarction within 6 months of cycle 1, day 1. [Subjects with a history of myocardial infarction between 6 and 12 months prior to cycle 1, day 1, who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event, may participate].
* Symptomatic coronary artery disease (CAD), e.g., angina Canadian Class II-IV. In any patient in whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present.
* An ECG recorded at screening showing evidence of cardiac ischemia (ST depression of ≥ 2 mm, measured from isoelectric line to the ST segment). If in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present.
* Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions and/or ejection fraction < 40% by multigated acquisition (MUGA) scan or < 50% by echocardiogram and/or magnetic resonance imaging (MRI);
* Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes.
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study medication.
* Patients requiring dual anti-platelets treatment for cardiac conditions or patients who are on anticoagulation for arterial or venous thrombosis. Patients with known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Patients that are pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through at least 30 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 2 years
  The estimated MTD would be the highest dose at which 0 out of 3 or 1 out of 6 subjects experience a dose-limiting toxicity (DLT), i.e. dose with an observed DLT rate of less than 0.33.

CONTACTS AND LOCATIONS:
Overall Officials: Changchun Deng, MD, PhD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No